CLINICAL TRIAL: NCT05522816
Title: A Phase 1, Dose Escalation Trial to Evaluate the Safety, Tolerability and Activity of Topical Administrations of Three Different Strengths of KX01 Ointment in Patients With Plaque Type Psoriasis
Brief Title: KX01 Ointment Phase 1 Study in Patients With Plaque Type Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B14-201
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2022-08

CONDITIONS: Psoriasis
Keywords: KX01; Ointment; Psoriasis; Phase I; Clinical trial
MeSH Terms: conditions — Psoriasis | interventions — tirbanibulin; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: The study will be sequentially performed in four stages, including stage 1 to stage 4. If no major safety concern was identified in the previous stage, as well as an unanimous consent by the sponsor and the principle investigator(s), the study will proceed to the next stage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and masking will be conducted in stage 1 and stage 2. Eight patients are randomized to received KX01 or placebo control in a ratio of 3:1 (KX01 versus placebo) in these 2 stages. Double blind are applied to the assignment of KX01 and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- KX01 0.01% in stage I (Experimental): Six patients in the stage 1 will receive KX01 0.01% (0.1 mg/g) for 2 weeks, followed by 1-week wash-out, another 2-week treatment, and then 2-week follow-up.
  Interventions: Drug: KX01 0.01% (0.1 mg/g)
- Placebo in stage 1 (Placebo Comparator): Two patients in the stage 1 will receive placebo treatment for 2 weeks, followed by 1-week wash-out, another 2-week treatment, and then 2-week follow-up.
  Interventions: Drug: Placebo
- KX01 0.1% in stage 2 (Experimental): Six patients in the stage 2 will receive KX01 0.1% (1.0 mg/g) for 4 weeks, followed by 2-week follow-up.
  Interventions: Drug: KX01 0.1% (1.0 mg/g)
- Placebo in stage 2 (Placebo Comparator): Two patients in the stage 2 will receive placebo treatment for 4 weeks, followed by 2-week follow-up.
  Interventions: Drug: Placebo
- KX01 1% for 5 days in stage 3 (Experimental): Six patients in stage 3 will receive 1% KX01 (10 mg/g) once daily for consecutive 5 days and then receive post-treatment follow-up on Day 6, 15 and 29.
  Interventions: Drug: KX01 1% (10 mg/g) for 5 days
- KX01 1% for consecutive 5 days and 2 days rest for 1 cycle, and repeat up to 4 cycles in stage 4 (Experimental): Six patients in stage 4 will be treated with daily KX01 1% (10 mg/g) ointment for consecutive 5 days and 2 days rest for 1 cycle, and repeat up to 4 cycles. And post-treatment follow-up visits will be conducted 14 days (Follow-up visit 1) and 28 days (Follow-up visit 2) after the end of cycle 4 treatment.
  Interventions: Drug: KX01 1% (10 mg/g) for consecutive 5 days and 2 days rest for 1 cycle, and repeat up to 4 cycles

INTERVENTIONS:
Drug: KX01 0.01% (0.1 mg/g) — Stage 1: 6 patients (KX01 0.01% [0.1 mg/g])
  Arms: KX01 0.01% in stage I
Drug: Placebo — Contains same excipients with KX01 but do not contain Tirbanibulin
  Arms: Placebo in stage 1; Placebo in stage 2
Drug: KX01 0.1% (1.0 mg/g) — Stage 2: 6 patients (KX01 0.1% [1.0 mg/g])
  Arms: KX01 0.1% in stage 2
Drug: KX01 1% (10 mg/g) for 5 days — Stage 3: 6 patients (KX01 1% [10 mg/g]) for 5 days
  Arms: KX01 1% for 5 days in stage 3
Drug: KX01 1% (10 mg/g) for consecutive 5 days and 2 days rest for 1 cycle, and repeat up to 4 cycles — Stage 4: 6 patients (KX01 1% [10 mg/g])for consecutive 5 days and 2 days rest for 1 cycle, and repeat up to 4 cycles
  Arms: KX01 1% for consecutive 5 days and 2 days rest for 1 cycle, and repeat up to 4 cycles in stage 4

SUMMARY:
This is a Phase I dose escalation study to assess the safety, tolerability and activity of three different strengths of topical KX01 in the treatment of patients with plaque-type psoriasis.

DETAILED DESCRIPTION:
This is a Phase I dose escalation study to assess the safety, tolerability and activity of three different strengths of topical KX01 (Tirbanibulin Ointment) in the treatment of patients with plaque-type psoriasis. The study will be performed in four stages as below.

Stage I: 6 patients (KX01 0.01% [0.1 mg/g]) + 2 patients (placebo); Stage II: 6 patients (KX01 0.1% [1.0 mg/g] + 2 patients (placebo); Stage III: 6 patients (KX01 1% [10 mg/g]) for 5 days; Stage IV: 6 patients (KX01 1% [10 mg/g]), duration escalation for up to 4 cycles.

If there's no major safety concern in the previous stage with an unanimous consent by the sponsor and the principle investigator, the study proceeded to the next stage.

The primary objective is to evaluate the safety and tolerability of three different strengths of KX01 ointment in patients with plaque-type psoriasis. The secondary objective is to gain evidence regarding the activity of three different strengths of KX01 ointment in patients with plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with plaque-type psoriasis, 20 years and older.
* Patient has a confirmed diagnosis of chronic plaque-type psoriasis for at least six months. For stage 4, PGA should be ≧3 &≦5 at baseline.
* A single lesion of ≥ 16 square centimetre and ≤ 625 square centimetre in size for Stage 1 and 2, and ≥ 16 square centimetre and ≤ 100 square centimetre in size for Stage 3 and 4 are selected as the target lesion (assessed at screening and Day 1).
* Medical history, vital signs, physical examination, standard 12-lead ECG and laboratory investigations have to be clinically insignificant or within laboratory reference ranges for the relevant laboratory tests, unless the investigator consider the deviation for out of range values to be irrelevant for the purpose of the study.
* No other disorders that, in the investigator's opinion, will prevent the patient from safely participating in this study or interfere with the evaluation of the patient's psoriasis.
* Patient is able to discontinue the use of any systemic medication or therapy for psoriasis.
* For females, either of the following conditions will be met: 1. Not of childbearing potential: Surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal; 2. Of childbearing potential: Negative serum pregnancy test at screening and not lactating, Either abstaining from sexual activity, or have to agree to use an accepted method of contraception, and agree to continue with the same method throughout the study.
* Male patients with partners of childbearing potential have to be willing to use contraception during the study and three months after end of treatment and is not to donate sperm for the duration of the study and for 3 months thereafter.
* Patient have to be able to provide written informed consent prior to the initiation of any study related procedures and able to comply with all the requirements of the study.

Exclusion Criteria:

* History of hypersensitivity to the investigational medicinal product (IMP) or to medicinal products with similar chemical structures.
* Presence of a skin disorder other than psoriasis in the target areas to be evaluated, including forms of inflammatory or non-inflammatory skin disorders that might interfere with determining efficacy or tolerability of the IMP.
* Severe forms of psoriasis or forms of psoriasis other than plaque psoriasis.
* All systemic psoriasis medications, including psoralens and ultraviolet A radiation treatments or other systemic immunosuppressive medication, are not allowed within five half-lives or 4 weeks (whichever is longer) prior to the first administration of the IMP.
* The use of topical therapies for psoriasis, including ultraviolet light B, on the target lesion to be studied within two weeks prior to the first administration of the IMP.
* Previous treatment with anti-tumor necrosis factor/interleukin (IL)-12/IL-23 or any other monoclonal antibodies within three months prior to the first administration of the IMP.
* Presence or history of any clinically significant acute or chronic disease which could interfere with the patient's participation or study outcome and at discretion of the clinical investigator.
* Patient with drug-induced psoriasis and is unable to discontinue the causal agent(s).
* Patient using prescription or non-prescription systemic drugs (e.g. vitamins and dietary, herbal supplements, paracetamol, aspirin or non-steroidal anti-inflammatory drugs [NSAIDs]) that might have an effect on psoriasis and is unable to maintain the stable dose or discontinue the dose during the study period.
* Participation in another study with an experimental drug, where the last administration of the previous IMP is within 4 weeks (or within five elimination half-lives for chemical entities or two elimination half-lives for antibodies or insulin, whichever is longer) before administration of IMP in this study, at the discretion of the investigator.
* A positive serum pregnancy test (beta human chorionic gonadotropin) or lactation.
* Vulnerable patients, e.g. persons in detention.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Adverse event at Stage 1 | Day 50
  Incidence of adverse event
Adverse event at Stage 2 | Day 43
  Incidence of adverse event
Adverse event at Stage 3 | Day 29
  Incidence of adverse event
Adverse event at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  Incidence of adverse event
Local tolerability score at Stage 1 | Day 50
  4-point (0-3) rating scale; higher scores mean a worse outcome
Local tolerability score at Stage 2 | Day 43
  4-point (0-3) rating scale; higher scores mean a worse outcome
Local tolerability score at Stage 3 | Day 29
  4-point (0-3) rating scale; higher scores mean a worse outcome
Local tolerability score at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  4-point (0-3) rating scale; higher scores mean a worse outcome
Vital signs at Stage 1 | Day 50
  any abnormal vital sign with clinical significance
Vital signs at Stage 2 | Day 43
  any abnormal vital sign with clinical significance
Vital signs at Stage 3 | Day 29
  any abnormal vital sign with clinical significance
Vital signs at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  any abnormal vital sign with clinical significance
12-lead ECG at Stage 1 | Day 36
  any abnormal finding of 12-lead ECG with clinical significance
12-lead ECG at Stage 2 | Day 29
  any abnormal finding of 12-lead ECG with clinical significance
12-lead ECG at Stage 3 | Day 29
  any abnormal finding of 12-lead ECG with clinical significance
12-lead ECG at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  any abnormal finding of 12-lead ECG with clinical significance
Hematology assessments at Stage 1 | Day 36
  any abnormal hematologic lab data with clinical significance
Clinical chemistry assessments at Stage 1 | Day 36
  any abnormal chemical lab data with clinical significance
Urinalysis assessments at Stage 1 | Day 36
  any abnormal urine lab data with clinically significant
Hematology assessments at Stage 2 | Day 29
  any abnormal hematologic lab data with clinical significance
Clinical chemistry assessments at Stage 2 | Day 29
  any abnormal chemical lab data with clinical significanc
Urinalysis assessments at Stage 2 | Day 29
  any abnormal urine lab data with clinically significant
Hematology assessments at Stage 3 | Day 29
  any abnormal hematologic lab data with clinical significance
Clinical chemistry assessments at Stage 3 | Day 29
  any abnormal chemical lab data with clinical significanc
Urinalysis assessments at Stage 3 | Day 29
  any abnormal urine lab data with clinically significant
Hematology assessments at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  any abnormal hematologic lab data with clinical significance
Clinical chemistry assessments at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  any abnormal chemical lab data with clinical significanc
Urinalysis assessments at Stage 4 | 28 days after the end of cycle 4 treatment (each cycle is 7 days)
  any abnormal urine lab data with clinically significant

SECONDARY OUTCOMES:
Change between baseline and end of treatment in target area score (TAS) at Stage 1 | Stage 1: Up to Day 36
  Change between baseline and end of treatment in TAS that evaluates the target lesion's erythema (0-4), plaque elevation (0-4) and scaling (0-4) on a five-point scale for each item (higher scores mean a worse outcome)
Change between baseline and end of TAS at Stage 2 | Up to Day 29
  Change between baseline and end of treatment in TAS that evaluates the target lesion's erythema (0-4), plaque elevation (0-4) and scaling (0-4) on a five-point scale for each item
Change between baseline and end of TAS at Stage 3 | Up to Day 6
  Change between baseline and end of treatment in TAS that evaluates the target lesion's erythema (0-4), plaque elevation (0-4) and scaling (0-4) on a five-point scale for each item
Change between baseline and end of TAS at Stage 4 | Up to the end of cycle 4 treatment (each cycle is 7 days)
  Change between baseline and end of treatment in TAS that evaluates the target lesion's erythema (0-4), plaque elevation (0-4) and scaling (0-4) on a five-point scale for each item
TAS 50 at Stage 1 | Up to Day 36
  ≧50% reduction in TAS score from baseline at the end of treatment
TAS 50 at Stage 2 | Up to Day 29
  ≧50% reduction in TAS score from baseline at the end of treatment
TAS 50 at Stage 3 | Up to Day 6
  ≧50% reduction in TAS score from baseline at the end of treatment
TAS 50 at Stage 4 | Up to the end of cycle 4 treatment (each cycle is 7 days)
  ≧50% reduction in TAS score from baseline at the end of treatment
Physician global assessment (PGA) score of the target lesion at the end of treatment of Stage 1 | Up to Day 36
  Achieving a score of "clear" (grade 0) or "almost clear" (grade 1) and at least 2 grade improvement from the baseline score in a 7-point score (0-6, higher scores mean a worse outcome).
PGA score of the target lesion at the end of treatment of Stage 2 | Up to Day 29
  Achieving a score of "clear" (grade 0) or "almost clear" (grade 1) and at least 2 grade improvement from the baseline score in a 7-point score
PGA score of the target lesion at the end of treatment of Stage 3 | Up to Day 6
  Achieving a score of "clear" (grade 0) or "almost clear" (grade 1) and at least 2 grade improvement from the baseline score in a 7-point score
PGA score of the target lesion at the end of treatment of Stage 4 | Up to the end of cycle 4 treatment (each cycle is 7 days)
  Achieving a score of "clear" (grade 0) or "almost clear" (grade 1) and at least 2 grade improvement from the baseline score in a 7-point score
Disease relapse at Stage 2 | Day 43
  Relapse is the loss of more than 50% of TAS improvement from baseline in patients who achieve a clinically meaningful response. Clinical meaningful response is defined as a reduction of ≥50% in TAS from baseline during the treatment.
Disease relapse at Stage 3 | Day 15 and Day 29
  Relapse is the loss of more than 50% of TAS improvement from baseline in patients who achieve a clinically meaningful response. Clinical meaningful response is defined as a reduction of ≥50% in TAS from baseline during the treatment.
Disease relapse at Stage 4 | 14 days after cycle 4 treatment and 28 days after cycle 4 treatment (each cycle is 7 days)
  Relapse is the loss of more than 50% of TAS improvement from baseline in patients who achieve a clinically meaningful response. Clinical meaningful response is defined as a reduction of ≥50% in TAS from baseline during the treatment.
Plasma KX01 concentrations (ng/ml) at Stage 1 | Up to Day 36
  Detection of plasma KX01 concentrations (ng/ml)
Plasma KX01 concentrations (ng/ml) at Stage 2 | Up to Day 29
  Detection of plasma KX01 concentrations (ng/ml)
Plasma KX01 concentrations (ng/ml) at Stage 3 | Up to Day 15
  Detection of plasma KX01 concentrations (ng/ml)
Plasma KX01 concentrations (ng/ml) at Stage 4 | 14 days after cycle 4 treatment (each cycle is 7 days)
  Detection of plasma KX01 concentrations (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Bon Hong, M.D., Principal Investigator — Department of Dermatology, National Taiwan University Hospital, Taipei, Taiwan; Po-Yuan Wu, M.D., Ph.D., Principal Investigator — Department of Dermatology, China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No